CLINICAL TRIAL: NCT03234673
Title: The Effect of Preceding Fractional Co2 Laser Either With Tacrolimus, Calcipotriol or With NB-UVB in the Treatment of Stable Generalized Vitiligo
Brief Title: The Effect of Fractional Co2 Laser Either With Tacrolimus, Calcipotriol or NB-UVB in Stable Generalized Vitiligo
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Mostafa Tawfik, clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEOPFCLEWTCOWNITTOSGV
Record Dates: First submitted 2017-07-27; First posted 2017-07-31 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Vitiligo Vulgaris
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Tacrolimus group): (Experimental): fractional CO2 laser therapy and Tacrolimus ointment 1
  Interventions: Drug: Tacrolimus ointment
- Group B (Calcipotriol group): (Experimental): fractional CO2 laser therapy and Calcipotriol ointment
  Interventions: Drug: calcipotriol ointment
- Group C (NB-UVB group): (Experimental): fractional CO2 laser therapy and NB-UVB twice weekly
  Interventions: Drug: NB-UVB

INTERVENTIONS:
Drug: Tacrolimus ointment — 3 sessions of fractional CO2 laser one month apart Patients will start treatment Tarolimus ointment twice daily for 3 months.
  Other Names: tarolimus ointment
  Arms: Group A (Tacrolimus group):
Drug: calcipotriol ointment — 3 sessions of fractional CO2 laser one month apart Patients will start treatment Calcipotriol ointment twice daily for 3 months.
  Other Names: calcipoheal
  Arms: Group B (Calcipotriol group):
Drug: NB-UVB — 3 sessions of fractional CO2 laser one month apart Patients will start treatment NB-UVB phototherapy twice weekly for 3 months
  Other Names: narrow band ultraviolet rays B
  Arms: Group C (NB-UVB group):

SUMMARY:
Vitiligo is an acquired disorder of the skin and mucous membranes characterized by well circumscribed depigmented macules and patches that occur secondary to selective destruction of melanocytes (Zhang et al., 2009).

Generalized vitiligo is the most common clinical presentation and often involves the face and acral regions (Alikhan et al., 2011).

DETAILED DESCRIPTION:
Combined vitiligo treatments have been found to be superior to monotherapies regarding efficacy, early response and safety (Kandaswamy et al., 2013).

Fractionated lasers represent a new modality for skin resurfacing based on the theory of fractional photothermolysis introduced by Manstein et al (2004). These lasers were shown to be efficient in treating facial photo aging changes as well as scars, and have an improved safety and recovery profile compared with traditional CO2 laser resurfacing. Fractionated lasers do not ablate the entire epidermis and thereafter leave intact skin between coagulated necrotic columns. This characteristic facilitates the skin healing process (Bogdan et al., 2010)

ELIGIBILITY:
Inclusion Criteria:

* patients with stable vitiligo
* nonsegmental vitiligo will be recruited
* A patient reporting no new lesions, no progression of existing lesions, and absence of Koebner phenomenon during the previous year

Exclusion Criteria:

1. Patients with active infection.
2. Reported histories of koebnerization.
3. History of keloid formation or hypertrophic scars.
4. Pregnant or lactating females.
5. Bleeding tendency.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
1- Re-pigmentation : that will be subjectively rated with a previously reported scoring system (Ghiya et al., 2016). | up to 3 months
  G0, < 25% repigmentation (poor)
  * G1, 25-50% repigmentation (fair)
  * G2, 50-75% repigmentation (good)
  * G3 > 75% repigmentation (excellent).

SECONDARY OUTCOMES:
The VASI percent change | every month for 3 months
  The VASI percent change will be calculated by subtracting the pre- procedure VASI score from the post-procedure VASI score and dividing by the pre-procedure VASI score.

OTHER OUTCOMES:
- Frequency and types of side effects. | 3 months
  pain, scarring, hyperpigmentation
- Patient satisfaction. The patient overall satisfaction will be assessed after 6 months according to Wong and Vasconez (2011). Overall satisfaction: | 3 months
  1. dissatisfied
  2. neutral
  3. somewhat satisfied
  4. moderately satisfied
  5. very satisfied

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ezzedine K, Eleftheriadou V, Whitton M, van Geel N. Vitiligo. Lancet. 2015 Jul 4;386(9988):74-84. doi: 10.1016/S0140-6736(14)60763-7. Epub 2015 Jan 15. PMID 25596811
- [Result] Kandaswamy S, Akhtar N, Ravindran S, Prabhu S, Shenoi SD. Phototherapy in Vitiligo: Assessing the Compliance, Response and Patient's Perception about Disease and Treatment. Indian J Dermatol. 2013 Jul;58(4):325. doi: 10.4103/0019-5154.113944. PMID 23919018
- [Result] Bogdan Allemann I, Kaufman J. Fractional photothermolysis--an update. Lasers Med Sci. 2010 Jan;25(1):137-44. doi: 10.1007/s10103-009-0734-8. PMID 19787413
- [Result] Wong L, Vasconez HC. Patient satisfaction after Nd:YAG laser-assisted lipolysis. Ann Plast Surg. 2011 May;66(5):561-3. doi: 10.1097/SAP.0b013e31820b3d1e. PMID 21451378